CLINICAL TRIAL: NCT06216951
Title: Evaluation of Post-operative Pain After Vital Pulpotomy in Molars With Symptomatic Pulpitis: A Prospective Clinical Study
Brief Title: Post-Operative Pain After Vital Pulpotomy in Molars With Symptomatic Pulpitis
Acronym: POPAVPT
Status: Completed | Type: Observational
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Hasibe Elif Kuru, Assistant Professor, Uşak University
Other Study IDs: 180-180-13
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Pulpitis; Post Operative Pain; Toothache
Keywords: toothache; pulpitis; pulpotomy; pain; postoperative
MeSH Terms: conditions — Pulpitis; Pain, Postoperative; Toothache; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with symptomatic pulpitis: vital permanent molars with symptomatic pulpitis in patients aged between 7-70
  Interventions: Procedure: Vital Pulpotomy

INTERVENTIONS:
Procedure: Vital Pulpotomy — Vital pulpotomy involves the removal of the coronal pulp, while MTA is used to seal the root orifices. It is clear that vital pulp treatments for symptomatic pulpitis are a more reliable, cost-effective, and generally easier option than root canal treatment (RCT) once the mineral trioxide aggregate (MTA) is introduced in dentistry. In vital pulpotomy, as opposed to RCT, tooth healing and symptoms are diminished while the vitality of the tooth is maintained. Furthermore, vital pulpotomy is a significantly more practical and economical treatment alternative than RCT.
  Other Names: vital pulp amputation

SUMMARY:
The goal of this clinical trial is to investigate post-operative pain (PEP) in teeth with symptomatic pulpitis following Vital Pulpotomy Treatments (VPT) with Calcium Silicate Cement (CSC). The main questions it aims to answer are:

* Is the post-operative pain one week after VPT significantly lower than pre-operative pain in permanent molars with symptomatic pulpitis?
* How does post-operative pain in these teeth correlate with patient-related factors, such as age, gender, and painkiller intake?

Participants will:

* Undergo Vital Pulpotomy Treatment with Calcium Silicate Cement (MTA)
* Provide pain level assessments before VPT, immediately post-treatment, and at 24, 72 hours, and 1 week after treatment.

If there is a comparison group:

Researchers will compare the post-operative pain levels in teeth with symptomatic pulpitis undergoing VPT to assess its effectiveness in reducing pain compared to a control group not undergoing the treatment.

DETAILED DESCRIPTION:
Informed Consent:

Volunteers or parents will receive detailed information about protocols, risks, and benefits. Informed consent was obtained in writing after providing subject information, and participants could withdraw voluntarily at any time.

Sample Size Calculation:

Sample size calculation, utilizing G. Power-3.1.9.2, aimed at relationship analyses with a 95% confidence level, α=0.05, effect size of 0.30, and theoretical power of 0.80, resulting in a minimum sample size of 108.

Treatment Procedure:

Vital pulpotomy, administered by experienced professionals, involved local anesthesia, rubber dam isolation, caries removal, pulp amputation, hemostasis, application of ProRoot MTA and glass ionomer, and permanent restoration. Pain scores, assessed using the modified Wong-Baker scale, were recorded pre-treatment, at 24 and 72 hours post-procedure, along with inquiries about painkiller usage.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 7 and 70 years
* The teeth with diagnosis of irreversible symptomatic pulpitis
* Permanent first and second molars with vital pulp
* PAI ≤ 2 with vital pulp. (Ørstavik D, Kerekes K, & Eriksen HM (1986) The periapical index: A scoring system for radiographic assessment of apical periodontitis Dent Traumatol 2(1) 20-34, https://doi.org/10.1111/j.1600-9657.1986.tb00119.x.)

Exclusion Criteria:

* Clinical or radiographic signs of a necrotic pulp
* The presence of a sinus, buccal tenderness, pathological mobility or evidence of pathology on a periapical radiograph
* Teeth with horizontal or vertical root fractures
* Swelling, acute endodontic, or periodontal abscess
* Insufficient tooth tissue for a restoration, teeth requiring a post
* Unable to give informed consent
* Contraindicated systemic disease
* Allergies the local anesthesia
* Antibiotics, biphosphonates, and corticosteroid intake during the 7 days before treatment.
* Pregnancy or breastfeeding.
* Patients who needed endodontic treatment on several teeth to avoid a potentially confused pain referral.

Ages: 7 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged between 7 and 70 with a noncontributory medical history presented for endodontic treatment at the Department of Endodontics and Department of Pediatric Dentistry, Faculty of Dentistry, Usak University, Turkey
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Assesment | 1) on treatment day, before starting the treatment; 2)24 hours later; 3)72 hours later and 4) 1 week later
  Pain scores before and after treatment will be assessed using a modified Wong-Baker pain rating scale. The patients and parents will be given with comprehensive information and instructed to indicate their level of pain using a pain rating scale (0 = no pain, 1 = slight pain, 2 = moderate pain, 3 = severe pain) before treatment, at 24 hours, and 72 hours after the procedure. Additionally, they will be asked about the use of painkillers.

CONTACTS AND LOCATIONS:
Overall Officials: Berk Çelikkol, Dr, Principal Investigator — Usak University School of Dentistry
Locations (1):
- Usak University School of Dentistry Department of Endodontics, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
due to possible plagiarism issues, we are kindly requesting that the study descriptions be shared only after journal publication

REFERENCES:
- [Background] Lin LM, Ricucci D, Saoud TM, Sigurdsson A, Kahler B. Vital pulp therapy of mature permanent teeth with irreversible pulpitis from the perspective of pulp biology. Aust Endod J. 2020 Apr;46(1):154-166. doi: 10.1111/aej.12392. Epub 2019 Dec 21. PMID 31865629
- [Background] Zanini M, Hennequin M, Cousson PY. A Review of Criteria for the Evaluation of Pulpotomy Outcomes in Mature Permanent Teeth. J Endod. 2016 Aug;42(8):1167-74. doi: 10.1016/j.joen.2016.05.008. Epub 2016 Jun 20. PMID 27339631
- [Background] Witherspoon DE, Small JC, Harris GZ. Mineral trioxide aggregate pulpotomies: a case series outcomes assessment. J Am Dent Assoc. 2006 May;137(5):610-8. doi: 10.14219/jada.archive.2006.0256. PMID 16739540
- See also: American Association of Endodontics, Clinical Guideline on Vital Pulp Therapy — https://www.aae.org/wp-content/uploads/2021/05/VitalPulpTherapyPositionStatement_v2.pdf